CLINICAL TRIAL: NCT02922127
Title: A Prospective, Randomized, Single-blind Study to Compare the Effects of Daily Ulipristal Acetate (UPA) 10mg With a Combined Oral Contraceptive (COC) Pill on Breast Epithelial Cell Proliferation in Reproductive Age Women
Brief Title: Compare Daily Ulipristal Acetate and Combined Oral Contraceptive Effects on Breast Epithelial Cell Proliferation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Weill Medical College of Cornell University (Other); Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Principal Investigator, Carolyn Westhoff, Professor, Department of Obstetrics and Gynecology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AAAQ8498
Record Dates: First submitted 2016-07-25; First posted 2016-10-04 (Estimated); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Contraception
Keywords: Ulipristal Acetate (UPA); Breast Cancer; Combined Oral Contraceptive (COC)
MeSH Terms: conditions — Breast Neoplasms | interventions — ulipristal acetate; Contraceptives, Oral, Combined; Ethinyl Estradiol-Norgestrel Combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ulipristal Acetate (Other): 20 women will randomized to daily use of 10mg of ulipristal acetate
  Interventions: Drug: Ulipristal Acetate
- Combined Oral Contraceptive (Other): 20 women will be randomized to daily use of a combined oral contraceptive pill
  Interventions: Drug: Combined Oral Contraceptive Pill

INTERVENTIONS:
Drug: Ulipristal Acetate — Daily use of Ulipristal Acetate
  Other Names: Ella
  Arms: Ulipristal Acetate
Drug: Combined Oral Contraceptive Pill — Daily use of Oral Contraceptive Pill
  Other Names: Portia
  Arms: Combined Oral Contraceptive

SUMMARY:
Breast cancer accounts for almost a quarter of all cancers in women. In the United States (U.S.) in 2014, more than 230,000 women were diagnosed and 40,000 died of breast cancer. There is an urgent need to develop acceptable means of preventing breast cancer both for high risk and average risk women.

The proposed study is a clinical trial in premenopausal women aged 18-39 to evaluate the capacity of daily Ulipristal Acetate (UPA) to reduce breast epithelial cell proliferation (increase in number of cells in the breast) and to measure its effect compared to that found with a combined estrogen-progestin oral contraceptive (COC). UPA is an anti-progestin in use as daily medication up to 12 months for the treatment of abnormally heavy bleeding at menstruation due to uterine fibroids, and is currently in trials in the U.S. to evaluate its use as a daily contraceptive.

The investigators will use breast biopsies to compare breast cell proliferation, comparing biopsies at the end of 3 months treatment to biopsies taken at baseline in the 2 groups (UPA and COC). The investigators will also compare the changes in the 2 groups to each other. The comparison of the effect of UPA to that of a conventional COC is because of UPA's potential use as a daily contraceptive.

Cell proliferation in the breast occurs throughout the menstrual cycle. The actions of hormones on the breast are rapid and an anti-progestin such as UPA, which will block the action of progesterone in the breast, would be predicted to quickly lower breast cell proliferation in premenopausal women. Effects of UPA on the uterus continue to be studied and are reassuring. COC use has not been found to lower breast cell proliferation and is not associated with any decrease in risk of breast cancer.

The changes in breast cell proliferation will also be compared to changes seen on breast MRI. If the changes are highly correlated future studies will be able to be done without the need for breast biopsies.

DETAILED DESCRIPTION:
This will be a randomized controlled parallel group clinical trial with blinded evaluation to be carried out at 2 academic medical centers: Columbia University Medical Center and Weill Cornell Medical College. The investigators will screen healthy women aged 18-39 who meet inclusion/exclusion criteria and will enroll them for the study.

After the informed consent process and study enrollment, study participation will begin with a baseline cycle. The main goal of the baseline cycle is to identify the occurrence and the timing of ovulation. Starting at about day 6 of the baseline cycle, participants will undergo blood sampling for progesterone (P4) levels at intervals of every 2-3 days. An increase of P4 to greater than 3 ng/mL, confirmed by a second such value, will indicate ovulation and eligibility to continue in the study. The participant's baseline breast MRI and biopsy (see below) will be scheduled to occur in the mid luteal phase, about 7 days after the first increase (>3 ng/mL) in P4. The investigators will randomly assign which breast has the first biopsy, and women will return for a post-biopsy visit about 7 days later. At the post-biopsy visit, the investigators will assess acceptability of the MRI and biopsy to the participants using visual analog scales (VAS) as well as interview.

At the beginning of the next menstrual period, women will begin the treatment phase of the study. They will receive random assignment to either UPA or COC at the study center and receive their first dose and a 4-week supply of study drug. During cycles 1 and 2 they will return to the study site every 2 weeks for assessment, blood draws and to receive the next cycle of study drug. During the third cycle, they will return to the study site twice weekly for more frequent testing and monitoring. Each cycle will be 28 days, corresponding to usual COC packaging. At day 75-77 of treatment women will undergo the second breast MRI, immediately followed by a biopsy of the contralateral breast to that biopsied at baseline. An end-of-study visit, including checking the incision site and a repeat assessment of acceptability of the MRI and biopsy to the participants, will occur about 7 days later. Participants will also be asked to rate their preference for an MRI versus a biopsy, were it possible to do a study with only one of these procedures.

Participants will have up to 24 study visits, and at each visit, participants will be asked about adverse events and use of any concomitant medications. Participants will have a high sensitivity urine pregnancy test at baseline and immediately preceding each MRI and preceding the first dose of study medication. Any participant with a positive pregnancy test will be immediately withdrawn from the study.

Breast Biopsies Breast biopsies will take place immediately following each breast MRI. Women will receive 24-hour telephone follow-up, and make a visit within one week following each breast biopsy to ensure that the biopsy site is healing without incident.

MRI For each participant, the baseline and follow-up MRI will be done using the same machine. Each MRI study will undergo an immediate wet read to assure adequate quality and to identify any unexpected pathology that would mandate clinical evaluation and withdrawal from the study. A limited report indicating technical adequacy and absence of major clinical abnormalities will be recorded in the patient record.

Breast MRI and breast biopsy visits will take place at the Center for Breast Imaging at Columbia University Medical Center.

ELIGIBILITY:
Inclusion Criteria:

1. Women between 18 and 39 years of age (inclusive).
2. In good health, with regular menstrual cycles between 21 and 35 days and with intra-individual variation of less than or equal to 5 days.
3. Volunteers who are postpartum or who aborted in the first or second trimester must have had two normal menstrual cycles (3 bleeding episodes) prior to screening.
4. No use of any other hormonal contraception within two normal menstrual cycles (3 bleeding episodes) prior to screening.
5. If previous use of injectable Depo Provera, subject must have had two normal menstrual cycles (3 bleeding episodes) prior to screening.
6. Not at risk for pregnancy:

   1. Using a copper intra uterine device (IUD), or
   2. Willing to protect all further acts of intercourse with condoms, or
   3. Not hetero-sexually active, or
   4. Having undergone previous tubal ligation, or
   5. Partner sterilized or vasectomized.
7. Body Mass Index (BMI) < 30 kg/m2 and not having previously undergone bariatric surgery.
8. Diastolic blood pressure (BP) ≤ 90 mm Hg and systolic BP ≤ 140 mm Hg after at least 5 minutes in a sitting position. Hypertensive subjects who are treatment controlled may obtain a waiver for participation.
9. Willing and able to follow all study requirements, including use of the study medication and willing to give information related to study medication use as required during the study, in the opinion of the investigator.
10. Able to give informed consent to participate in the study.

Exclusion Criteria:

1. Currently pregnant as confirmed by positive high-sensitivity urine pregnancy test.
2. Currently breast-feeding or within 30 days of discontinuing breast feeding at screening.
3. Undiagnosed abnormal genital bleeding.
4. Known hypersensitivity to an active substance or any of the excipients of the study treatments.
5. Abnormal clinical breast examination at screening.
6. Suspected hyperplasia or carcinoma of the endometrium.
7. Ovarian cyst > 25 mm observed on transvaginal or transabdominal ultrasound performed on the first visit of the Baseline cycle.
8. History of any diagnostic or therapeutic breast biopsy
9. Any of the known contraindications to COC use:

   1. History of or existing breast cancer, or other hormone sensitive neoplasia, or
   2. History of or current ischemic heart disease or stroke, or
   3. History of or current deep venous thrombosis or pulmonary embolism, or
   4. Systemic lupus erythematosus with positive or unknown antiphospholipid antibodies, or
   5. History of or current benign or malignant liver tumor, or
   6. Severe (decompensated) cirrhosis.
   7. Headaches with focal neurological symptoms.
10. Hereditary galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption.
11. Known or suspected alcoholism or drug abuse.
12. Known human immunodeficiency virus (HIV) infection.
13. Smoking 15 cigarettes or more per day, if in the opinion of the investigator or medically qualified designee, this would increase the risk for cardiovascular disease and thromboembolism based on risk factors.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2016-12-16 (Actual); Primary Completion 2019-10-21 (Actual); Study Completion 2019-10-21 (Actual)

PRIMARY OUTCOMES:
Change in breast epithelial cell proliferation rate | Baseline, three months
  The breast biopsies will be analyzed (measured by Ki67) at end of study treatment, as compared with baseline before initiation of treatment.

SECONDARY OUTCOMES:
Change in breast epithelial cell proliferation rate in the UPA group compared to the change in the COC group | Three months
  The breast biopsies will be analyzed (measured by Ki67).
Proportion of subjects using UPA who experience a categorical decrease in breast background parenchymal enhancement (BPE) | Baseline, three months
  This will be measured with contrast MRI.
Proportion of subjects experiencing a categorical decrease in breast BPE in the UPA group compared to the change in the COC group | Three months
  This will be measured with contrast MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Westhoff, MD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Columbia University Irving Medical Center, New York, New York
  - Weill Cornell Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Westhoff CL, Guo H, Wang Z, Hibshoosh H, Polaneczky M, Pike MC, Ha R. The progesterone-receptor modulator, ulipristal acetate, drastically lowers breast cell proliferation. Breast Cancer Res Treat. 2022 Apr;192(2):321-329. doi: 10.1007/s10549-021-06503-1. Epub 2022 Jan 11. PMID 35015210